CLINICAL TRIAL: NCT06522074
Title: Evaluating the Role of IGF-1 and S-Klotho in Plaque Phenotype and Vulnerability: The VISION Study
Acronym: VISION
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6347
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Heart Disease; Chronic Coronary Syndrome; Optical Coherence Tomography (OCT)
MeSH Terms: conditions — Myocardial Ischemia | interventions — Coronary Angiography; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coronary angiography with OCT — Intravascular imaging with Optical Coherence Tomography (OCT) in patients with chronic coronary syndrome who have been indicated for coronary angiographic will be used at the operator's discretion, for diagnostic purposes and/or to guide possible coronary artery disease treatment.

SUMMARY:
Insulin-like growth factor 1 (IGF-1) is the primary peripheral mediator of growth hormone (GH) and has pleiotropic effects on development, differentiation, metabolism, and cell survival. Several in vivo and in vitro studies suggest that IGF-1 may have a protective effect on atherosclerosis as it suppresses macrophage recruitment and activation, cytokine production, and extracellular matrix degradation while promoting smooth muscle cell migration and proliferation and extracellular matrix deposition. The protein sKlotho appears to be closely related to the GH-IGF-1 axis, and some animal and in vitro studies hypothesize its protective role in the cardiovascular system. The GH-IGF-1 axis and sKlotho influence mechanisms determining coronary atherosclerosis. Circulating levels of IGF-1 and sKlotho may correlate with the morphology of atherosclerotic plaques and particularly with the vulnerability of coronary lesions.

Objectives: To evaluate the correlation between atherosclerotic plaque phenotype and the GH-IGF-1 axis and sKlotho in patients with chronic coronary syndrome using intravascular imaging with Optical Coherence Tomography (OCT).

Methods:All patients with chronic coronary syndrome who meet the inclusion and exclusion criteria and undergo coronary angiography and intravascular imaging with optical coherence tomography will be included. At the end of the procedure, a blood sample will be taken to measure IGF-1, sKlotho, and GH receptor (GHR) polymorphism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic coronary syndrome undergoing coronary angiographic study.
* Patients undergoing intravascular imaging with OCT during coronary angiographic study at the operator's discretion, for diagnostic purposes and/or to guide possible coronary artery disease treatment.
* Patients with at least 18 years of age.
* Patients able to provide informed consent.

Exclusion Criteria:

* Pregnancy.
* Pathological excess or deficiency of IGF-1.
* Stage IV chronic renal failure.
* Severe liver disease.
* Cachexia and/or malnutrition states.
* BMI <18.5.
* HbA1C ≥ 8.5%.
* Left Ventricle Ejection Fraction (LVEF) <= 35%
* Patients with aorto-coronary bypass.
* OCT analysis conducted on vessels with previous percutaneous coronary intervention with stent implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with chronic coronary syndrome indicated for coronary angiographic study and who will undergo intravascular imaging with OCT, used at the operator's discretion, for diagnostic purposes and/or to guide possible coronary artery disease treatment.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between atherosclerotic plaque phenotype and plasma levels of IGF-1 and sKlotho protein and GH receptor (GHR) polymorphism | 2 years
  To assess the correlation between atherosclerotic plaque phenotype and plasma levels of IGF-1, sKlotho protein, and GH receptor (GHR) gene expression through intravascular imaging with Optical Coherence Tomography (OCT).

SECONDARY OUTCOMES:
correlation between atherosclerotic plaque phenotype and plasma levels of other hormones and inflammation markers | 2 years
  To assess the correlation between atherosclerotic plaque phenotype and plasma levels of thyroid-stimulating hormone (TSH), triiodothyronine (FT3), thyroxine (FT4), cortisol, adrenocorticotropic hormone (ACTH), follicle-stimulating hormone (FSH), luteinizing hormone (LH), estradiol, testosterone, inflammation markers (interleukin 6, C-reactive protein), vitamin D, and FGF-23 (fibroblast growth factor).

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Burzotta, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Cardiologia, Roma, Italy